CLINICAL TRIAL: NCT05376163
Title: Validity and Reliability of the Turkish Version of The Henry Ford Hospital Headache Disability Index (HDI) in Patients With Cervicogenic Headache
Brief Title: Validity of Headache Disability Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Prof.Dr., Hacettepe University
Other Study IDs: GO 22/670
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Neck Pain; Headache; Cervical Pain
Keywords: Cervicogenic headache; Cervical Spine; Validity
MeSH Terms: conditions — Neck Pain; Headache; Post-Traumatic Headache | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with headache: Individuals with headaches caused by neck problems
  Interventions: Other: Survey Study

INTERVENTIONS:
Other: Survey Study — Headache Disabilty Index (HDI) will be applied.

SUMMARY:
The aim of our study is to investigate the Turkish validity and reliability of The Henry Ford Hospital Headache Disability Questionnaire (HDI), which has not been previously studied in a Turkish version for any headache type in patients with cervicogenic headache.

DETAILED DESCRIPTION:
Headache is a health problem that is reported to occur in 66% of the global population, reducing both quality of life and work productivity. The most common type is tension headache with a prevalence of 38%, followed by migraine headaches with 10%. The incidence of cervicogenic ligament pain has been shown to be between 2.5 and 4.1%. It has been reported that although the prevalence of cervicogenic headache is low compared to tension-type headache and migraine, it affects the quality of life in patients similarly.he International Headache Society has defined cervicogenic headache as pain felt in at least one area of the face or head that radiates from a source in the neck. The most common clinical picture of cervicogenic headache is neck pain, which is usually unilateral and may radiate from the occipital region to the orbit. It has been suggested that neck pain and headache are common comorbidities. Cote et al. reported that headache complaint is 10 times more common in people with neck pain than in people without neck pain.It has been reported that an average of 60-80% of individuals suffering from chronic neck pain have headache problems. C.The validity and reliability studies of the questionnaire on headache in Turkey were generally conducted in patients with migraine. Dikmen et al. performed the Turkish validity and reliability study of the Headache Impact Test-6 (Headache Impact Test-6) questionnaire in patients with migraine. Ertaş et al. published the Turkish version of the Migraine Disability (MIDAS) Questionnaire in the same patient group. However, we could not find a Turkish validity and reliability study of a questionnaire in patients with cervicogenic headache in our country.

The Henry Ford Hospital Headache Disability Questionnaire (HDI), developed by Jacobson et al. in 1994, is a 25-item questionnaire that examines the effects of headache on daily life. This questionnaire has a two-factor structure emotionally and functionally. Scoring (No: 0, Sometimes:2, Yes:4) varies between 0 and 100. The higher the score, the more headache disability.

ELIGIBILITY:
Inclusion Criteria:

* Getting over 4 points from the Neck Disability Index
* According to the 3rd edition of the International Headache Disorders Classification System (International Headache Disorders Classification 3rd edition),having at least two of the following parameters, Development of headache temporally related to the onset of cervical problems Significant reduction of headache in parallel with the improvement of cervical problems Variation in headache severity with cervical region movements Decreased range of motion in the cervical region in addition to headache

Exclusion Criteria:

* Being diagnosed by a neurologist from any of the diagnoses of migraine, cluster headache syndrome, tension headache, chronic post-traumatic headache, drug-induced headache (ICD Diagnostic Codes).
* Having a history of any neurological or systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with cervicogenic headache.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Headache Disability Index (HDI) | 15 minutes
  Headache Disability Index evaluates the effects of headache on quality of life and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Onan, MSc, Study Chair — Hacettepe University; Özlem Ülger, Study Director — Hacettepe Üniversity
Locations (1):
- Hasan Erkan Kilinç, Ankara, Turkey (Türkiye)